CLINICAL TRIAL: NCT06267313
Title: Attention Training for COVID-19 Related Distress
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting participants
Sponsor: Palo Alto University (Other)
Responsible Party: Principal Investigator, Mikael Rubin, Assistant Professor, Palo Alto University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-078-PAU
Record Dates: First submitted 2024-02-17; First posted 2024-02-20 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Bias Modification (Experimental)
  Interventions: Behavioral: Attention Bias Modification
- Attention Control Training (Active Comparator)
  Interventions: Behavioral: Attention Control Training
- Neutral Training (Placebo Comparator)
  Interventions: Behavioral: Neutral training

INTERVENTIONS:
Behavioral: Attention Bias Modification — Training attention away from threat
  Arms: Attention Bias Modification
Behavioral: Attention Control Training — Training attention control
  Arms: Attention Control Training
Behavioral: Neutral training — Attention training with Neutral stimuli
  Arms: Neutral Training

SUMMARY:
The study aims to test whether attention training (attention bias modification or attention control training) reduces distress or COVID-19 related anxiety compared to a neutral condition.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 Anxiety Syndrome Scale > 7 and/or COVID-19 related loss

Exclusion Criteria:

* Does not speak English Fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
COVID-19 Anxiety Syndrome Scale | 0 days
  The measure is scored using a 5-point time anchored scale (0 = Not at all to 4 = Nearly every day over the last 2 weeks) and scores range between 0 and 20, with higher scores reflecting worse outcome.
COVID-19 Anxiety Syndrome Scale | 21 days
  The measure is scored using a 5-point time anchored scale (0 = Not at all to 4 = Nearly every day over the last 2 weeks) and scores range between 0 and 20, with higher scores reflecting worse outcome.
COVID-19 Anxiety Syndrome Scale | 49 days
  The measure is scored using a 5-point time anchored scale (0 = Not at all to 4 = Nearly every day over the last 2 weeks) and scores range between 0 and 20, with higher scores reflecting worse outcome.
COVID-19 Anxiety Syndrome Scale | 105 days
  The measure is scored using a 5-point time anchored scale (0 = Not at all to 4 = Nearly every day over the last 2 weeks) and scores range between 0 and 20, with higher scores reflecting worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available with accompanying manuscript
Supporting Information: Analytic Code
Time Frame: Analytic code will be shared with accompanying manuscript